CLINICAL TRIAL: NCT03327831
Title: UCI 14-92 / HS#2015-1889: Phase IV Study of Daylight Photodynamic Therapy With Aminolevulinic Acid for Actinic Keratoses
Brief Title: Study of Daylight Photodynamic Therapy With Aminolevulinic Acid for Actinic Keratoses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Christopher Zachary, Principal Investigator, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20151889
Record Dates: First submitted 2015-10-23; First posted 2017-10-31 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Actinic Keratosis
Keywords: aminolevulinic acid; pdt; photodynamic therapy; Photochemotherapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aminolevulinic Acid with daylight photodynamic therapy arm (Experimental): This study has a single, open label treatment arm. Patients will have topical aminolevulinic acid applied to the actinic keratoses in the treatment area (face/scalp) and will spend 2 hours outdoors in the shade to activate the medication. The patient then follow up in clinic 3 months and 6 months after their treatment to have the number of actinic keratoses counted.
  Interventions: Drug: Aminolevulinic Acid

INTERVENTIONS:
Drug: Aminolevulinic Acid — Topical application followed by activation by ambient sunlight
  Other Names: Kerastick

SUMMARY:
Photodynamic therapy is an effective treatment for actinic keratoses. In the United States topical aminolevulinic acid (ALA) is approved as a photosensitizing agent for this treatment, and it has traditionally been activated with the use of an in-office artificial light source. This clinical trial seeks to measure the safety and efficacy of using natural sunlight to activate the ALA.

DETAILED DESCRIPTION:
* Initial Visit:

  * study inclusion criteria reviewed
  * consent forms reviewed
  * creation of facial map for actinic keratoses
  * face cleansed with chlorhexidine soap
  * light curettage of precancerous skin lesions
  * application of topical aminolevulinic acid (ALA)
  * application of sunscreen
  * patient then spends 2 hours outdoors in a shaded area
  * after treatment the patient is to remain indoors for 48 hours
* 3 month follow up visit

  - facial map of actinic keratoses used to document treatment response
* 6 month follow up visit

  * facial map of actinic keratoses used to document treatment response

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of >10 actinic keratoses on head and neck
* Age ≥ 18 years (Because no dosing or adverse event data are currently available on the use of topical aminolevulinic acid in patients <18 years of age, children are excluded from this study)
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients currently undergoing anti-neoplastic therapy including but not limited to the following:

  * Topical imiquimod
  * Topical 5-fluorouracil
  * Topical ingenol mebutate
  * Topical diclofenac
  * Topical retinoids
  * Oral acitretin
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to aminolevulinic acid
* Patients with a known photosensitivity disorder including but not limited to porphyria, lupus, polymorphous light eruption, or immunobullous disease.
* Patients taking known photosensitizing medications including but not limited to griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, sulfonamides and tetracyclines.
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B Zachary, MBBS. FRC[, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aminolevulinic Acid With Daylight Photodynamic Therapy Arm
Started | 30
Completed | 28
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Aminolevulinic Acid With Daylight Photodynamic Therapy Arm
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 23
Age, Continuous [Mean (Full Range); unit: years] | 68.5 [50 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30
Actinic keratoses [Mean (Full Range); unit: Actinic keratoses] | 36.4 [11 to 105]
Average ambient lux [Mean (Full Range); unit: lux] — Ambient lux, or a measure of luminous flux per unit area from sunlight, is measured during treatment and will be analyzed to determine it if contributes to treatment efficacy. Patients measure their lux with a handheld luxometer (Suncheck Instruments, Model HS1010 Sun Nuclear Corporation, Melbourne).
  lux | 8,244 [2,000 to 16,820]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Number of Actinic Keratoses
Description: Percent change in number of actinic keratoses at 6 months
Time Frame: 0 (baseline) and 6 months
Measure: Median (Full Range); unit: % change in number of actinic keratoses
Units Other Than Participants: actinic keratosis
Arm/Group | Aminolevulinic Acid With Daylight Photodynamic Therapy Arm
Number analyzed (Participants) | 30
Number analyzed (actinic keratosis) | 105
% change in number of actinic keratoses | -75 [-92 to -35]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with adverse events such as crusting, erythema, edema, or pain
Time Frame: 2 days
Measure: Number; unit: participants
Arm/Group | Aminolevulinic Acid With Daylight Photodynamic Therapy Arm
Number analyzed (Participants) | 30
participants | 3

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Aminolevulinic Acid With Daylight Photodynamic Therapy Arm
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aminolevulinic Acid With Daylight Photodynamic Therapy Arm (N=30)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) — Pruritus of the skin
Pustules (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03327831/Prot_SAP_000.pdf